CLINICAL TRIAL: NCT06465745
Title: AltaValve Pivotal Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: 4C Medical Technologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5472
Record Dates: First submitted 2024-06-05; First posted 2024-06-20 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-03

CONDITIONS: Mitral Regurgitation; Mitral Insufficiency; Mitral Valve Incompetence; Mitral Valve Regurgitation; Mitral Incompetence
Keywords: Mitral Regurgitation; TMVR; Functional Regurgitation; Degenerative Regurgitation; Transcatheter Mitral Valve Replacement; Primary Regurgitation; Secondary Regurgitation
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Primary Cohort (Experimental): Designed to evaluate the safety and performance of the AltaValve System for the treatment of moderate-to-severe or severe MR in a targeted patient population without at least moderate mitral annular calcification (MAC).
  Interventions: Device: AltaValve System.
- Mitral Annular Calcification Cohort (MAC) (Experimental): Designed to evaluate the safety and performance of the AltaValve System for the treatment of moderate-to-severe or severe MR in a targeted patient population with moderate to severe MAC.
  Interventions: Device: AltaValve System.

INTERVENTIONS:
Device: AltaValve System. — Transcatheter Mitral Valve Replacement.

SUMMARY:
This is a prospective, single arm, multicenter, clinical trial designed to evaluate the safety and performance of the AltaValve System for the treatment of mitral regurgitation in a targeted patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Symptomatic New York Heart Association (NYHA) class II-IV.
* Moderate-to-severe or severe MR (3+) despite optimal guideline-directed medical therapy (GDMT) as determined by an independent Echo Core Lab.
* Unsuitable for surgery and Transcatheter Edge-toEdge Repair (TEER) as determined by the local site Heart Team.

Exclusion Criteria (Abbreviated List):

* Inability to understand the trial or a history of non-compliance with medical advice.
* Inability to provide signed Informed Consent Form (ICF).
* History of any cognitive or mental health status that would interfere with participation in the trial.
* Currently enrolled in any other pre-approval investigational trial (does not apply to long-term post-market trials unless these trials might clinically interfere with the current trial endpoints (e.g., limit use of trial-required medication, etc.)).
* Female subjects who are pregnant or planning to become pregnant within the trial period.
* Known hypersensitivity or contraindication to heparin, or warfarin without adequate alternative medications.
* Known hypersensitivity to nitinol (i.e., nickel allergy) that cannot be adequately medicated.
* Known hypersensitivity to contrast media that cannot be adequately medicated.
* Evidence of current left ventricular ejection fraction (LVEF) ≤ 25%.
* Concurrent medical condition with a life expectancy of less than 12 months.
* Transcatheter aortic repair or replacement within 90 days prior to the index procedure.
* Percutaneous coronary intervention (PCI) within 90 days prior to the index procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or heart failure hospitalization. | 12 months.

SECONDARY OUTCOMES:
All-cause mortality, disabling stroke, acute kidney injury (stage 3 or with renal replacement), mitral valve re-intervention (surgical or transcatheter), major bleeding requiring intervention. | 30 Days or hospital discharge (whichever is longer).
  Composite.
Technical success. | Day 0.
  Technical success will be considered achieve when all of the following are present:
  * Successful application of the delivery system as intended.
  * Successful device placement.
  * Reduction in mitral regurgitation grade to ≤ 2+.
Mitral valve re-intervention. | At 30 days, 6 months, 1 year, and annually thereafter for up to 5 years.
  Mitral valve re-intervention after index procedure
Changes in Kansas City Cardiomyopathy Questionnaire (KCCQ). | 6 months and 1 year.
  Quality of life improvement.
Changes in Six-minute walk test (6MWT). | 6 months and 1 year.
  Quality of life improvement.
New pacemaker rate. | 1 month, 6 months and 1 year.

CONTACTS AND LOCATIONS:
Locations (29):
- United States (20):
  - Abrazo Arizona Heart Hospital, Phoenix, Arizona
  - Dignity Health; St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - TMC Healthcare, Tucson, Arizona
  - Sutter Bay Hospitals, San Francisco, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Cardiovascular Institute of the South, Houma, Louisiana
  - MedStar Health Research Institute, Inc., Columbia, Maryland
  - William Beaumont Hospital, Royal Oak, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - AHS Hospital Corp., Morristown, New Jersey
  - New York Presbyterian Hospital-Columbia University Medical Center, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - The Charlotte-Mecklenburg Hospital; Atrium Health, Charlotte, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - South Oklahoma Heart Research, LLC., Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Germany (4):
  - Universitatsklinikum Bonn, Bonn
  - University Hospital Cologne - Heart Center, Cologne
  - Cardiac Research GmbH; St.-Johannes-Hospital Dortmund, Dortmund
  - Heart Center Trier, Trier
- Greece (2):
  - Onassis Cardiac Surgery Center, Athens
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
- Spain (3):
  - Hospital Clinic de Barcelona, Barcelona
  - Fundación para la investigación biomédica del hospital clínico San Carlos, Madrid
  - Hospital Álvaro Cunqueiro, Vigo